CLINICAL TRIAL: NCT04110314
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal- RCT #2
Brief Title: Patient Portal Reminder/Recall for Influenza Vaccination in a Health System- RCT 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01AI135029 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Vaccination; Reminder recall; Patient Portal
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Gain-framed portal reminders + Pre-commitment Prompts (Active Comparator): Participants receive gain-framed reminder/recall messages regarding influenza vaccination via the patient portal and a pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Gain-framed; Behavioral: Pre-commitment prompt
- Gain-framed portal reminders + No pre-commitment prompt (Active Comparator): Participants receive gain-framed reminder/recall messages regarding influenza vaccination via the patient portal and no pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Gain-framed
- Loss-framed portal reminders + Pre-commitment prompt (Active Comparator): Participants receive loss-framed reminder/recall messages regarding influenza vaccination via the patient portal and a pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Loss-framed; Behavioral: Pre-commitment prompt
- Loss-framed portal reminders + No pre-commitment prompt (Active Comparator): Participants receive loss-framed reminder/recall messages regarding influenza vaccination via the patient portal and a no pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Loss-framed
- No portal reminder + Pre-commitment prompt (Active Comparator): Participants do not receive any reminder/recall messages regarding influenza vaccination via the patient portal but do receive a pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season
  Interventions: Behavioral: Pre-commitment prompt
- No portal reminders + No pre-commitment prompt (No Intervention): Participants do not receive any reminder/recall messages regarding influenza vaccination via the patient portal and do not receive a pre-commitment prompt asking if they plan to receive the influenza vaccine in the upcoming season

INTERVENTIONS:
Behavioral: Portal Reminders for Influenza Vaccination: Gain-framed — Patients receive gain-framed reminder/recall messages via the patient portal to get an influenza vaccination.
  Arms: Gain-framed portal reminders + No pre-commitment prompt; Gain-framed portal reminders + Pre-commitment Prompts
Behavioral: Portal Reminders for Influenza Vaccination: Loss-framed — Patients receive loss-framed reminder/recall messages via the patient portal to get an influenza vaccination.
  Arms: Loss-framed portal reminders + No pre-commitment prompt; Loss-framed portal reminders + Pre-commitment prompt
Behavioral: Pre-commitment prompt — Patients receive a pre-commitment prompt asking about their intention to get an influenza vaccination
  Arms: Gain-framed portal reminders + Pre-commitment Prompts; Loss-framed portal reminders + Pre-commitment prompt; No portal reminder + Pre-commitment prompt

SUMMARY:
This trial is taking place in Los Angeles, CA among patients from primary care practices within the UCLA Health System.

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low. The investigators will assess the effectiveness of message-framing (gain-framed, loss-framed messages, no messages), as well as the effectiveness of a pre-commitment prompt (pre-commitment prompt, no prompt) asking about a patient's intention to get the influenza vaccination, using a 3 x 2 factorial design.

DETAILED DESCRIPTION:
Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices to not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients.

There has been considerable research on how best to communicate about vaccines with families. A number of studies have examined the impact of gain-framed (messages emphasizing the benefits of vaccination) versus loss-framed (messages emphasizing the risks of not getting vaccinated); however, the findings have been inconsistent across studies and by sub-population.

In addition to framing, another potential influence on the decision to vaccinate is pre-commitment. Previous studies suggest that, upon being prompted, indicating an intention to do something increases the likelihood of following through. Therefore, a pre-commitment prompt is being asked of half the participants in each arm to evaluate its impact on influenza vaccination.

The purpose of this randomized controlled trial is to evaluate the impact of gain-framed and loss-framed reminder-recall messages sent via the patient portal, pre-commitment prompts sent via the patient portal, and the interactions between the two type of messages and pre-commitment on influenza vaccination among UCLA Health System's primary care patients aged 6 months and older.

The proposed design of this randomized-controlled trial is a 3 x 2 factorial design.

Standard of care control (no reminder messages, no pre-commitment prompt) No portal messages, pre-commitment prompt Gain-framed portal messages, pre-commitment prompt Gain-framed portal messages, no pre-commitment prompt Loss-framed portal messages, pre-commitment prompt Loss-framed portal messages, no pre-commitment prompt

Hyp 1. Vaccination rates will differ by receipt of no reminders, gain-framed reminders and loss-framed reminders.

1a. Vaccination rates will be higher among patients receiving gain-framed reminders than among patients receiving no reminders.

1b. Vaccination rates will be higher among patients receiving loss-framed reminders than among patients receiving no reminders.

1c. Vaccination rates will be higher among patients receiving gain-framed reminders than among patients receiving loss-framed reminders.

Hyp 2. Vaccination rates will be higher among patients receiving a pre-commitment prompt than among patients not receiving any prompt.

For relevant study arms, the first R/R messages will be sent in October 2019.

ELIGIBILITY:
Inclusion Criteria:

* A patient within the UCLA Health System identified as a primary care patient per an internal algorithm,

Exclusion Criteria:

* A patient within the UCLA Health System not identified as a primary care patient per an internal algorithm

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430636 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Szilagyi, MPH, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California LA, Los Angeles, California, United States

REFERENCES:
- [Derived] Szilagyi PG, Albertin CS, Casillas A, Valderrama R, Duru OK, Ong MK, Vangala S, Tseng CH, Humiston SG, Evans S, Sloyan M, Bogard JE, Fox CR, Lerner C. Effect of Personalized Messages Sent by a Health System's Patient Portal on Influenza Vaccination Rates: a Randomized Clinical Trial. J Gen Intern Med. 2022 Feb;37(3):615-623. doi: 10.1007/s11606-021-07023-w. Epub 2021 Sep 1. PMID 34472020
- [Derived] Lerner C, Albertin C, Casillas A, Duru OK, Ong MK, Vangala S, Humiston S, Evans S, Sloyan M, Fox CR, Bogard JE, Friedman S, Szilagyi PG. Patient Portal Reminders for Pediatric Influenza Vaccinations: A Randomized Clinical Trial. Pediatrics. 2021 Aug;148(2):e2020048413. doi: 10.1542/peds.2020-048413. PMID 34321338

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gain-framed Portal Reminders + Pre-commitment Prompts | Gain-framed Portal Reminders + No Pre-commitment Prompt | Loss-framed Portal Reminders + Pre-commitment Prompt | Loss-framed Portal Reminders + No Pre-commitment Prompt | No Portal Reminder + Pre-commitment Prompt | No Portal Reminders + No Pre-commitment Prompt
Started | 71781 | 71492 | 72177 | 71512 | 71536 | 72138
Patients Who Met Inclusion | 36526 | 36388 | 36541 | 36377 | 36289 | 36411
Completed | 36526 | 36388 | 36541 | 36377 | 36289 | 36411
Not Completed | 35255 | 35104 | 35636 | 35135 | 35247 | 35727
Not completed — Did not meet inclusion criteria | 35255 | 35104 | 35636 | 35135 | 35247 | 35727

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gain-framed Portal Reminders + Pre-commitment Prompts | Gain-framed Portal Reminders + No Pre-commitment Prompt | Loss-framed Portal Reminders + Pre-commitment Prompt | Loss-framed Portal Reminders + No Pre-commitment Prompt | No Portal Reminder + Pre-commitment Prompt | No Portal Reminders + No Pre-commitment Prompt | Total
Number analyzed (Participants) | 36526 | 36388 | 36541 | 36377 | 36289 | 36411 | 218532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3686 | 3632 | 3727 | 3610 | 3655 | 3736 | 22046
  Between 18 and 65 years | 26288 | 26191 | 26265 | 26170 | 26180 | 26077 | 157171
  >=65 years | 6552 | 6565 | 6549 | 6597 | 6454 | 6598 | 39315
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female Female | 21088 | 20881 | 21058 | 21057 | 20947 | 20835 | 125866
  Male | 15437 | 15506 | 15482 | 15319 | 15342 | 15575 | 92661
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown | 1 | 1 | 0 | 1 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20096 | 20133 | 20115 | 20056 | 20401 | 20401 | 121202
  Black/African American | 1674 | 1666 | 1657 | 1649 | 1727 | 1533 | 9906
  Asian | 3867 | 3789 | 3886 | 3900 | 3715 | 3828 | 22985
  Other/Unknown | 10889 | 10800 | 10883 | 10772 | 10815 | 10649 | 64808
Region of Enrollment [Number; unit: participants]
  United States | 36526 | 36388 | 36541 | 36377 | 36289 | 36411 | 218532
Insurance Type [Count of Participants; unit: Participants]
  Private | 31307 | 31164 | 31302 | 31129 | 31148 | 31167 | 187217
  Public | 4642 | 4646 | 4671 | 4690 | 4584 | 4675 | 27908
  Other/UNK | 577 | 578 | 568 | 558 | 557 | 569 | 3407
Adults with diabetes [Count of Participants; unit: Participants] | 3660 | 3644 | 3663 | 3485 | 3534 | 3539 | 21525

OUTCOME MEASURES:

1. Primary Outcome: Receipt of the Annual Influenza Vaccine Among Index Patients.
Description: Receipt of the annual influenza vaccination (between 10/2/19 - 4/1/20) among index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  Index patients will be randomly selected individuals within an included household, eligible for the following groups (<18, 18-64 non-diabetic, 65+ non-diabetic, and 18+ diabetic). One index patient per group may be selected from each household.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/19, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Population: Each row represents a combination of intervention conditions in our factorial design. Each column represents patient subpopulations which received different versions of the intervention. The number analyzed in each cell is the number from that column's subpopulation assigned to that row's intervention combination.
Measure: Count of Participants; unit: Participants
Groups:
- Young Adults 18-64yr Without Diabetes: Participants ages 18-64 Without Diabetes
- Older Adults Greater Than or Equal to 65 yr Without Diabetes: Older adults with diabetes greater than or equal to 65 years without diabetes.
- Adults 18years or Older With Diabetes: Adults 18 years or older with Diabetes
- Children <18y: Participants age <18
Arm/Group | Young Adults 18-64yr Without Diabetes | Older Adults Greater Than or Equal to 65 yr Without Diabetes | Adults 18years or Older With Diabetes | Children <18y
Number analyzed (Participants) | 145166 | 29795 | 21525 | 22046
Participants
  No reminders and no pre-commitment: number analyzed (Participants) | 24133 | 5003 | 3539 | 3736
  No reminders and no pre-commitment | 8804 | 2795 | 2163 | 2123
  Loss-framed reminders and no pre-commitment: number analyzed (Participants) | 24246 | 5036 | 3485 | 3610
  Loss-framed reminders and no pre-commitment | 8880 | 2752 | 2077 | 2056
  Gain-frame reminders and no pre-commitment: number analyzed (Participants) | 24130 | 4982 | 3644 | 3632
  Gain-frame reminders and no pre-commitment | 8796 | 2772 | 2183 | 2076
  No reminders and pre-commitment: number analyzed (Participants) | 24200 | 4900 | 3534 | 3655
  No reminders and pre-commitment | 8937 | 2757 | 2144 | 2084
  Loss-frame reminders and pre-commitment: number analyzed (Participants) | 24210 | 4941 | 3663 | 3727
  Loss-frame reminders and pre-commitment | 9055 | 2753 | 2220 | 2203
  Gain-frame reminders and pre-commitment: number analyzed (Participants) | 24247 | 4933 | 3660 | 3686
  Gain-frame reminders and pre-commitment | 8883 | 2741 | 2249 | 2168
Statistical Analysis 1: Comparison: Young Adults 18-64yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [1.00 to 1.03] — These results compare the arm receiving a pre-commitment prompt to the arm receiving no pre-commitment prompt
Statistical Analysis 2: Comparison: Older Adults Greater Than or Equal to 65 yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.01] — These results compare the arm receiving a pre-commitment prompt to the arm receiving no pre-commitment prompt
Statistical Analysis 3: Comparison: Adults 18years or Older With Diabetes; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.99 to 1.03] — These results compare the arm receiving a pre-commitment prompt to the arm receiving no pre-commitment prompt
Statistical Analysis 4: Comparison: Children <18y; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.04] — These results compare the arm receiving a pre-commitment prompt to the arm receiving no pre-commitment prompt
Statistical Analysis 5: Comparison: Young Adults 18-64yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.98 to 1.01] — These results compare the arm receiving gain-framed reminders to the arm receiving no reminders
Statistical Analysis 6: Comparison: Older Adults Greater Than or Equal to 65 yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 0.99, 0.95% CI 2-sided [0.97 to 1.02] — These results compare the arm receiving gain-framed reminders to the arm receiving no reminders
Statistical Analysis 7: Comparison: Adults 18years or Older With Diabetes; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.97 to 1.01] — These results compare the arm receiving gain-framed reminders to the arm receiving no reminders
Statistical Analysis 8: Comparison: Children <18y; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.98 to 1.05] — These results compare the arm receiving gain-framed reminders to the arm receiving no reminders
Statistical Analysis 9: Comparison: Young Adults 18-64yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.99 to 1.02] — These results compare the arm receiving loss-framed reminders to the arm receiving no reminders
Statistical Analysis 10: Comparison: Older Adults Greater Than or Equal to 65 yr Without Diabetes; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.98 to 1.02] — These results compare the arm receiving loss-framed reminders to the arm receiving no reminders
Statistical Analysis 11: Comparison: Adults 18years or Older With Diabetes; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.97 to 1.02] — These results compare the arm receiving loss-framed reminders to the arm receiving no reminders
Statistical Analysis 12: Comparison: Children <18y; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.04] — These results compare the arm receiving loss-framed reminders to the arm receiving no reminders

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events.
Description: We did not collect adverse event information. We monitored whether reminder recall through the portal was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Gain-framed Portal Reminders + Pre-commitment Prompts | Gain-framed Portal Reminders + No Pre-commitment Prompt | Loss-framed Portal Reminders + Pre-commitment Prompt | Loss-framed Portal Reminders + No Pre-commitment Prompt | No Portal Reminder + Pre-commitment Prompt | No Portal Reminders + No Pre-commitment Prompt
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT04110314/Prot_SAP_000.pdf